CLINICAL TRIAL: NCT06589492
Title: A Cross-sectional Study on the Comparison of Serum SIRT-1 and MMP-9 Levels of Patients With Bronchiectasis and Healthy Controls
Brief Title: Comparison of Serum SIRT-1 and MMP-9 Levels of Patients With Bronchiectasis and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Dilara Ulger Ozbek, principal investigator, Cumhuriyet University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Biochemistry AD
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bronchiectasis Adult
Keywords: Bronchiectasis; MMP-9; SIRT-1
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT scan (No Intervention): Chest high-resolution CT scan will be performed for diagnosis of patients.
- Age, gender (No Intervention): Age and gender information of patients will be obtained for comparison.
- Measurement of MMP-9 and SIRT-1 levels in blood serum (Experimental): It involves taking 5ml of blood from participants to measure mmp-9 and SIRT-1 levels in blood serum.
  Interventions: Diagnostic Test: Measurement of MMP-9 and SIRT-1 levels in blood serum

INTERVENTIONS:
Diagnostic Test: Measurement of MMP-9 and SIRT-1 levels in blood serum — Measurement of MMP-9 and SIRT-1 levels in blood serum, Collection of 5 ml Blood samples
  Arms: Measurement of MMP-9 and SIRT-1 levels in blood serum

SUMMARY:
The purpose of this a cross-sectinol study is to measure the levels of MMP-9 and SIRT-1 levels in patients with bronchiectasis and healthy controls. The aim is to compare the serum levels of these molecules between patients and controls.

* Is the MMP-9 level increasing or decreasing?
* Is the SIRT-1 level increasing or decreasing in patients?
* Is the disease related to age and gender? Participants will only have one 5 ml blood sample drawn when they visit the chest illness clinic. Molecule levels will be measured in this blood's serum.

The patient group participants will be scanned once with high-resolution chest CT.

Apart from this, comparisons will be made using the age and gender information of the participants.

DETAILED DESCRIPTION:
In the overall study population of 60 subjects who applied to the Sivas Cumhuriyet University Faculty of Medicine Research and Practice Hospital Chest Diseases Clinic. The study population was selected regardless of age and gender. Participants selected bronchiectasis patients (n=30) who had symptoms (cough, sputum production) and had their diagnosis confirmed by a chest high-resolution CT scan within the previous year. The study excluded individuals with bronchiectasis not associated with cystic fibrosis and who had a worsening episode (according to the 2017 European Respiratory Society expert consensus criteria) (16) or had taken antibiotics during the previous four weeks. The study enrolled healthy controls (n=30) through advertisements who had acceptable chest X-ray and spirometry results and no lower airway symptoms or serious systemic disorders. The study eliminated individuals who were pregnant or nursing, as well as those with low comprehension. SIRT-1 and MMP-9 levels in the serum of the study group were determined by the ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis patients who were symptoms (cough, sputum production)
* Individuals whose diagnosis was confirmed by a high-resolution chest CT scan taken within the previous year

Exclusion Criteria:

* Individuals with bronchiectasis associated with cystic fibrosis and who had a worsening episode
* individuals who were pregnant or nursing
* those with low comprehension
* taken antibiotics during the previous four weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
MMP-9 and SIRT-1 levels (ng/mL) mesurment in the blood serum to compare between patient and control. | not measured in time frame. general (1. day)
  MMP-9 and SIRT-1 levels mesured in the blood serum. The most common side effect when blood is taken from the patient is slight bruising and swelling in the arm due to needle sticking. There will be no other serious side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet University, Sivas, Si̇vas Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
can be published after being converted into a working article